CLINICAL TRIAL: NCT00308321
Title: Long Term Tapering or Standard Steroids for Nephrotic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: Tracy Assari, Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03NU13
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: long term tapering of prednisolone — 60mg/m2/day (0-4 weeks); 60mg/m2 alternate days (5-6 weeks); 50mg/m2 alternate days (week 7-8); 40mg/m2 alternate days (week 9-10); 30mg/m2 alternate days (week 11-12); 20mg/m2 alternate days (week 13-14); 10mg/m2 alternate days (week 15-16)
Drug: standard prednisolone treatment — 60mg/m2/day week 0-4; 40mg/m2 on alternate days week 5-8

SUMMARY:
Parallel group double blind randomised in patients with first episode corticosteroid sensitive nephrotic syndrome comparing time to relapse and adverse effects associated with a longer tapering steroid regimen with standard regime

ELIGIBILITY:
Inclusion Criteria:

* newly presenting nephrotic syndrome, urine albumin/protein creatinine ratio >200mg/mmol on early morning urine sample, hypoalbuminemia (<25g/L)

Exclusion Criteria:

* prior treatment with steroids or cytotoxic agents underlying systemic disorder or exposure to agents known to be associated with newly presenting steroid sensitive nephrotic syndrome

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2003-09; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Time to first relapse | 5 months
Assessment of steroid induced morbidity | 5 months

SECONDARY OUTCOMES:
frequent relapsing and steroid dependant disease | 5 months
Time to relapse | 5 months
serious adverse events | 5 months
use of other immunosuppressive agents | 5 months
Achenbach child behaviour checklist | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Trompeter, Principal Investigator — Great Ormond Street Hospital; Peter Houtman, Principal Investigator — Children's Hospital, Leicester
Locations (1):
- Institute of Child Health, London, United Kingdom

REFERENCES:
- [Derived] Hahn D, Samuel SM, Willis NS, Craig JC, Hodson EM. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD001533. doi: 10.1002/14651858.CD001533.pub7. PMID 39171624